CLINICAL TRIAL: NCT00450528
Title: The Kinetics of D-Dimers After Abdominal Surgery as a Function of the Invasiveness of Surgery
Brief Title: Kinetics of D-Dimers After Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Other Study IDs: StV 31-2006
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Last update posted 2007-10-24 (Estimated); Status verified 2007-10

CONDITIONS: Natural Kicetics of d-Dimers After Surgery
Keywords: D-dimers; surgery; kinetics

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the natural kinetics of D-dimers that occur after abdominal surgery.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a potentially fatal disease with an estimated incidence of 0.1%. One third of the VTE occur as pulmonal embolism with a mortality up to 25% (White RH. Circulation 107:2003)

Serum d-dimer levels are used as sensitive marker for the diagnosis of VTE (Kelly J et al. Arch Intern Med, 162: 2002). Because of its sensitivity, the determination of serum D-dimer levels is an accepted method to exclude VTE in the outpatient setting meaning that VTE may be excluded in case of normal D-dimer levels (Kelly J. Lancet 359: 2002). The specificity of the D-dimer testing, however, is low. This is true especially in the postoperative phase. The interpretation of elevated D-dimer levels in surgical patients remains elusive.

The natural kinetics of D-dimers after surgery is not known. The question to what extent D-dimer levels rise after surgery and how long it may take D-dimer levels to return to normal after surgery is not yet determined. This information is needed to be able to use D-dimer testing for VTE diagnosis in surgical patients.

In this study, D-dimer levels are measured in surgical patients immediately before (day 0) and repeatedly after surgery. D-dimer level measurement will be stopped after D-dimer levels returned to normal.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective surgery

Exclusion Criteria:

* age < 18 years
* patients not speaking german
* patients involved in another study
* pregnancy
* concommitant inflammatory disease
* patients with oral anticoagulation
* patients having received fresh frozen plasma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-02; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dindo, MD, Principal Investigator — University of Zurich
Locations (1):
- Univeryity Hospital, Clinic for Visceral- and Transplantation Surgery, Zurich, Canton of Zurich, Switzerland